CLINICAL TRIAL: NCT06109935
Title: A Multi-centre, Prospective, Open Label, Single-arm, Non-interventional Post-marketing Study to Investigate the Long-term Safety and Clinical Parameters of Sogroya® Treatment in Children With Short Stature Due to Growth Hormone Deficiency Where Epiphysial Discs Are Not Closed Under Normal Clinical Practice Conditions in Japan Special Use-results Surveillance on Long Term Use of Sogroya® in Children With Short Stature Due to Growth Hormone Deficiency (GHD) Where Epiphysial Discs Are Not Closed
Brief Title: Special Use-results Surveillance on Long Term Use of Sogroya® in Children With Short Stature Due to Growth Hormone Deficiency Where Epiphysial Discs Are Not Closed
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-5005; U1111-1274-4223 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Growth Hormone Deficiency in Children
MeSH Terms: interventions — somapacitan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with GHD: Participants will be treated with commercially available Sogroya® according to routine clinical practice at the discretion of the treating physician. Administration will be according to the approved product labelling. The decision to treat a participant with Sogroya® is made at the treating physician's discretion before and independently from the decision to include the patient in this study.
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — Sogroya® treatment regimen will be in accordance with the approved product labelling in Japan.
  Other Names: Sogroya®

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Sogroya® in children with short stature due to growth hormone deficiency where epiphysial discs are not closed under real-world clinical practice in Japan. The study will last for about 1 year (at shortest) to 3 years (at longest) depending on when the participant takes part in the study. The participant will be asked to answer questionnaire(s) about how they feel about the growth hormone (GH) product treatment once during the study (at about 3 months after starting the Sogroya® treatment) and about 3 months after starting the Sogroya® treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. The decision to initiate treatment with commercially available Sogroya® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study. Both GH treatment naïve and non-naïve children are eligible.
3. Male or female age 0 to 18 years (exclusive) at the time of signing informed consent.
4. Diagnosis with short stature due to GHD where epiphysial discs are not closed according to local normal clinical practice.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Treatment with any investigational drug within 30 days prior to baseline (the starting date of Sogroya® treatment).
3. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
4. Contraindication described in approved product labelling in Japan.

   1. Patients with hypersensitivity to the active substance or to any of the excipients
   2. Patients with malignant tumour
   3. Female patients who are either pregnant or likely to be pregnant

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with short stature due to Growth Hormone Deficiency (GHD) where epiphysial discs are not closed under normal clinical practice conditions in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse reactions (AR) | From baseline (week 0) to end of study (up to 156 weeks)
  Measured as count of reactions.

SECONDARY OUTCOMES:
Number of adverse events (AEs) | From baseline (week 0) to end of study (up to 156 weeks)
  Measured as count of events.
Number of serious adverse events (SAEs) | From baseline (week 0) to end of study (up to 156 weeks)
  Measured as count of events.
Number of serious adverse reactions (SARs) | From baseline (week 0) to end of study (up to 156 weeks)
  Measured as count of reactions.
Change in height velocity (HV) | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
  Measured in centimeter (cm)/year.
Change in bone age | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
  Measured in years.
Change in ratio of bone age/chronological age | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
Change in height standard deviation score (HSDS) | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
Change in height velocity standard deviation score (HVSDS) | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
Change in insulin-like growth factor-I standard deviation score (IGF-I SDS) | Every 12 months from baseline (week 0) to end of study (up to 156 weeks)
  Measured as score ranging from -10 to +10. Negative scores indicated a IGF-I below the mean IGF-I for a child with the same age and gender, whereas positive scores indicated a IGF-I above the mean IGF-I for a child with the same age and gender. For participants with low IGF-I SDS at baseline, a positive change from baseline in IGF-I SDS indicated a better outcome.
Growth hormone device assessment tool (G-DAT) | At 12 weeks
  Measured as count of patients choosing the individual response category. G-DAT is a questionnaire to gather information on how they feel about the GH product device assessed as "very easy", "easy", "neither difficult or easy", "difficult" or "very difficult" where "very easy" is best and "very difficult" is worst.
Growth hormone patient preference questionnaire (GH-PPQ) | At 12 weeks
  Measured as count of patients choosing the individual response category. GH-PPQ is a disease specific questionnaire which measures the patient's growth hormone treatment preference.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (84):
- Japan (84):
  - Hoshigaoka Seicho Clinic_Pediatrics, Aichi
  - Iwayama Pediatric_Pediatrics, Aichi
  - Asai Clinic_Pediatrics, Aichi
  - Mutsu general hospital, Aomori
  - Asahikawa Medical Univ. Hospital_Pediatrics, Asahikawa, Hokkaido
  - Beppu Medical Center, Beppu-shi, Oita-ken
  - Inomata Child Clinic_Pediatrics, Chiba
  - Seirei Sakura Citizen Hospital_Pediatrics, Chiba
  - Kurume University Hospital, Pediatrics, Fukuoka
  - Fukuoka University Hospital, Fukuoka-shi, Fukuoka-ken
  - Kyushu University Hospital, Fukuoka-shi, Fukuoka
  - Gifu University Hospital, Gifu
  - Ota Memorial Hospital_Pediatrics, Gunma
  - Kato Clinic, Hachioji-shi, Tokyo-to
  - Hamamatsu University Hospital, Hamamatsu-shi, Shizuoka
  - Hello Clinic, Higashimatsuyama-shi, Saitama-ken
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyogo-ken
  - Yonekura Child Clinic_Pediatrics, Hiroshima
  - Hyogo prefectural kobe children's hospital, Hyōgo
  - Nakasako Kids Clinic_Pediatrics, Hyōgo
  - Nagai Kids Clinic_Pediatrics, Hyōgo
  - Sunsun Kodomo Clinic, Ichikawa-shi, Chiba-ken
  - Komatsu Municipal Hospital_Pediatrics, Ishikawa
  - Fukushima Seishi Ryougoen, Iwaki-shi, Fukushima-ken
  - Shimane University Hospital_Pediatrics, Izumo-shi, Shimane-ken
  - Kagoshima University hospital_Pediatrics, Kagoshima
  - University Hospital Kyoto Prefectual University of Medicine, Kamigyo-ku, Kyoto
  - Muza Kawasaki Pediatric Clinic_Pediatrics, Kanagawa
  - Oguchi Higashi Hospital_Pediatrics, Kanagawa
  - Hanamaru Kids Clinic_Pediatrics, Kanagawa
  - Odawara Municipal Hospital_Diabetes and Endocrinology, Kanagawa
  - Nippon Medical School Musashikosugi Hospital_Neurological Surgery, Kawasaki-shi, Kanagawa-ken
  - Hospital of the University of Occupational And Environmental Health Japan, Pediatrics, Kitakyusyu-shi, Fukuoka
  - Mominoki Hospital, Pediatrics, Kochi-shi, Kochi
  - Kumamoto University Hospital, Pediatrics, Kumamoto-shi, Kumamoto
  - Ayabe City Hospital, Kyoto
  - University of Miyazaki Hospital_Pediatrics, Miyazaki
  - Haga Red Cross Hospital, Moka-shi, Tochigi-ken
  - Kodomohamirai Morioka Kodomo Clinic, Morioka-shi, Iwate-ken
  - Aichi Medical University Hospital, Nagakute-shi, Aichi
  - Ina Central Hospital_Nagano, Nagano
  - Nagasaki University Hospital_Pediatrics, Nagasaki
  - Nagoya City University Hospital, Pediatric, Nagoya, Aichi
  - Naha City Hospital, Naha-shi, Okinawa
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa-ken
  - Nara Medical University Hospital_Pediatrics, Nara
  - Nara Prefecture General Medical Center, Nara-shi, Nara
  - Niigata University Medical & Dental Hospital_Pediatrics, Niigata-shi, Niigata
  - Hyogo Medical University Hospital_Pediatrics, Nishinomiya-shi, Hyogo-ken
  - Iwate Medical University Hospital, Numakunai
  - Aichi Children's Health and Medical Center, Obu-shi, Aichi
  - Okayama University Hospital_Pediatrics, Okayama
  - Asahigawasou Ryouiku Iryou Center_Pediatrics, Okayama
  - Chibana Clinic, Okinawa
  - Osaka City General Hospital_Endocrinology and Diabetes Mellitus, Osaka
  - Kibounomori Clinic, Osaka
  - JCHO Osaka Hospital_Pediatric, Osaka
  - Saiseikai Suita Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Yasuhara Children's Clinic, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - Kojiya Kodomo clinic, Ota-ku, Tokyo-to
  - Okubo Kids Clinic, Ozu-shi, Ehime-ken
  - Clinic for Children and Youths_Pediatrics, Saitama
  - Sakai Smile Kids Clinic, Sashima-gun, Ibaraki-ken
  - JR Sendai Hospital, Sendai-shi, Miyagi-ken
  - Shiga university of Medical Science Hospital_Pediatrics, Shiga
  - Shiga General Hospital_Diabetes and Endocrinology, Shiga
  - My Clinic Ohkubo, Shizuoka
  - Shizuoka Saiseikai General Hospital_Pediatrics, Shizuoka
  - Hamamatsu Medical Center, Shizuoka
  - Iwata City Hospital_Pediatrics, Shizuoka
  - Shizuoka Children's Hospital, Department of Diabetes and metabolism, Shizuoka-shi, Shizuoka
  - Sakura Kids Clinic_Pediatrics, Tokyo
  - National Center for Child Health and Dev, Endo and Metabo, Tokyo
  - Tanaka Growth Clinic, Tokyo
  - Akiruno Clinic_Pediatrics, Tokyo
  - Ehime University Hospital, Toon-shi, Ehime
  - Murakami Pediatric and Allergy clinic, Toyama-shi, Toyama-ken
  - Fujita Health University Hospital, Pediatrics, Toyoake, Aichi
  - Toyohashi Municipal Hospital, Toyohashi-shi, Aichi-ken
  - Tendo City Hospital_Pediatrics, Yamagata
  - Ikeda Pediatrics Clinic, Yamagata-shi, Yamagata-ken
  - Yamaguchi University Hospital_Pediatrics, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com